CLINICAL TRIAL: NCT00487019
Title: Comparative Study of Two Antibiotic Regimen - Penicillin G/Gentamicin Versus Ampicillin/Gentamicin in Empirical Treatment of Early Onset Neonatal Septicaemia
Brief Title: Management of Early Onset Neonatal Septicaemia: Selection of Optimal Antibacterial Regimen for Empiric Treatment
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Collaborators: Estonian Science Foundation (Other Government); European Society for Paediatric Infectious Diseases (Other)
Other Study IDs: 038FAR042005
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Early Onset Neonatal Sepsis
Keywords: ampicillin; penicillin G; gentamicin; neonatal sepsis; empiric therapy
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Neonates aged <72 h and needing antibacterial therapy for early onset neonatal sepsis
- 2: Same as group 1

SUMMARY:
A prospective two-center antibiotic regimen switch study will be conducted to compare the clinical efficacy of two antibiotic regimens - penicillin/gentamicin versus ampicillin/gentamicin - in the empirical treatment of early onset neonatal sepsis. The influence of either regimen on bowel colonization pattern and on the development of antibiotic resistance of gut microflora will also be assessed. The primary endpoint is the need for a change in antibacterial treatment within 72 hours of therapy, based on pre-defined criteria. Secondary endpoints will be the incidence rate and etiology of early and late onset neonatal sepsis and susceptibility pattern of causative microorganisms; mortality rate within 60 days; duration of hospitalization in NICU; duration of artificial ventilation; colonization pattern and susceptibility of colonizing bacteria (including resistance to empiric antibiotic regimen).

DETAILED DESCRIPTION:
A prospective randomized two-centre antibiotic regimen switch study will be conducted in the NICU-s of Tartu University Clinics and of Tallinn Children's Hospital. Initially all patients who need empiric treatment for early onset neonatal sepsis (as defined by Schrag et al. 2002) in Tartu will be treated with penicillin/gentamicin and those in Tallinn with ampicillin/gentamicin. When half of the needed subjects have been recruited, departmental antibiotic regimen will be switched so that ampicillin is used in Tartu and penicillin in Tallinn. Based on the present patient population and hospitalization rate, about 120-150 babies, eligible for the study will be admitted to either units every a year.

In all subjects predefined pre- and intranatal risk factors of infection will be registered. During the NICU stay laboratory and clinical signs of infection, need for respiratory support and vasoactive therapy, enteral and parenteral nutrition will be recorded.

Blood, CSF and urine cultures will be taken according to the routine of the ward but certainly before every change in antibacterial treatment. For colonization studies nasopharyngeal or tracheal and anal swabs will be collected from all neonates admitted during the study period on admission and thereafter biweekly until discharge from the NICU or until the 60th day of treatment. A separate protocol will be followed for microbiological investigations.

The endpoints:

The primary endpoint is the need for a change in antibacterial treatment within 72 hours. In discussions with clinical experts in both wards the following criteria for the change in antibacterial treatment were defined:

1. proven or suspected meningitis or abdominal infection
2. isolation from a relevant site of the mother or an infant of a microorganism, resistant to initial empiric treatment regimen in babies with early onset neonatal sepsis or septic shock
3. deterioration of the clinical status on initial antibiotic regimen and suspected/proven neonatal sepsis
4. suspected/proven late onset sepsis or nosocomial infection (defined as the development of clinical/ laboratory signs of infection at postnatal age of 72 hours or more)
5. other situations, where the treating physician considers change in antibiotic regimen necessary - the reasons will be recorded in the case report form Patients, who die before 72 hours or in whom the antibacterial therapy is changed for other than the above-mentioned reasons, will be handled as treatment failures.

Secondary endpoints will be the following:

* incidence rate and etiology of early and late onset neonatal sepsis, susceptibility pattern of causative microorganisms
* incidence rate and etiology of nosocomial sepsis, susceptibility pattern of causative microorganisms
* mortality rate within 60 days
* duration of hospitalization in NICU stay
* duration of artificial ventilation
* colonization pattern and susceptibility of colonizing bacteria (including resistance to empiric antibiotic regimen).

ELIGIBILITY:
Inclusion Criteria:

* All neonates, admitted to the study NICU-s at the age of less than 72 hours and needing early empiric antibiotic treatment according to pre-defined criteria as described by Schrag et al. (2002)

Exclusion Criteria:

* Subjects, who on clinical or other indications (e.g. suspected/proven meningitis or abdominal cavity infection, isolation of resistant bacteria from the mother of a neonate with severe sepsis) need antibiotic treatment other than specified in the study protocol and infants who are likely to be transferred to other units within 24 hours.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates hospitalised within 72h of life and requiring empirical antibacterial treatment for early onset neonatal sepsis.
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2006-08; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irja Lutsar, MD, PhD, Study Chair — University of Tartu
Locations (2):
- Estonia (2):
  - Tallinń's Childrens Hospital, Paediatric Intensive Care Unit, Tallinn
  - Tartu University Clinics, Department of Paediatric Intensive Care, Tartu

REFERENCES:
- [Background] Schrag S, Gorwitz R, Fultz-Butts K, Schuchat A. Prevention of perinatal group B streptococcal disease. Revised guidelines from CDC. MMWR Recomm Rep. 2002 Aug 16;51(RR-11):1-22. PMID 12211284